CLINICAL TRIAL: NCT01305551
Title: Bioequivalence Study of the Fixed Dose Combination of 5 mg Saxagliptin and 500 mg Metformin Hydrochloride (HCl) XR Tablet Relative to a 5 mg Saxagliptin (Onglyza™) Tablet and a 500 mg Metformin HCl XR (Glifage® XR Marketed in Brazil by Merck S.A.) Tablet Co-Administered to Healthy Subjects in the Fasted and Fed States
Brief Title: BE Study of the Fixed Dose Combination of 5 mg Saxagliptin and 500 mg Metformin HCl XR Tablet Relative to a 5 mg Saxagliptin (Onglyza™) Tablet and a 500 mg Metformin HCl XR (Glifage® XR Marketed in Brazil by Merck S.A.) Tablet Co-Administered to Healthy Subjects in the Fasted and Fed States
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: CV181-146
Record Dates: First submitted 2011-02-25; First posted 2011-02-28 (Estimated); Last update posted 2014-06-05 (Estimated); Status verified 2014-06

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — saxagliptin; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment A-Saxagliptin+Metformin XR (Experimental): 5mg Saxagliptin + 500 mg Metformin XR Tablets, once on Day 1 only, administered together in the fasted state.
  Interventions: Drug: Saxagliptin; Drug: Metformin XR
- Treatment B-Saxagliptin/Metformin XR FDC (Experimental): 5mg Saxagliptin / 500 mg Metformin XR FDC tablet, once on Day 1 only, administered in the fasted state.
  Interventions: Drug: Saxagliptin/Metformin XR FDC
- Treatment C-Saxagliptin+Metformin XR (Experimental): 5mg Saxagliptin + 500 mg Metformin XR Tablets, once on Day 1 only, administered together in the fed state.
  Interventions: Drug: Saxagliptin; Drug: Metformin XR
- Treatment D-Saxagliptin/Metformin XR FDC (Experimental): 5mg Saxagliptin / 500 mg Metformin XR FDC tablet, once on Day 1 only, administered in the fed state.
  Interventions: Drug: Saxagliptin/Metformin XR FDC

INTERVENTIONS:
Drug: Saxagliptin — Tablet, Oral, 5 mg, once on Day 1 only
  Other Names: Onglyza
  Arms: Treatment A-Saxagliptin+Metformin XR; Treatment C-Saxagliptin+Metformin XR
Drug: Metformin XR — Tablet, Oral, 500 mg, once on Day 1 only
  Other Names: Glifage XR
  Arms: Treatment A-Saxagliptin+Metformin XR; Treatment C-Saxagliptin+Metformin XR
Drug: Saxagliptin/Metformin XR FDC — Tablet, Oral, 5/500 mg, once on Day 1 only
  Other Names: Onglyza/Glucophage
  Arms: Treatment B-Saxagliptin/Metformin XR FDC; Treatment D-Saxagliptin/Metformin XR FDC

SUMMARY:
The purpose of this study is to demonstrate the bioequivalence (BE) of Saxagliptin and Metformin from a 5 mg Saxagliptin/500 mg Metformin extended release (XR) fixed dose combination (FDC) tablet relative to 5 mg Onglyza™ and 500 mg Glifage® XR (marketed in Brazil by Merck S.A.) tablets administered together in both the fasted and fed states.

DETAILED DESCRIPTION:
Primary purpose: To demonstrate the bioequivalence of Saxagliptin and Metformin from a 5 mg Saxagliptin/500 mg Metformin XR FDC tablet relative to 5 mg Onglyza™ and 500 mg Glifage® XR (marketed in Brazil by Merck S.A.) tablets administered together in both the fasted and fed states.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* Women of childbearing potential (WOCBP) who are using acceptable method of contraception
* Women who are not nursing

Exclusion Criteria:

* History of Gastrointestinal (GI) disease
* Any GI surgery that could impact study drug absorption
* History of allergy to drug class or related compounds
* History of allergy to metformin or other similar acting agents.
* History of any significant drug allergy.
* Estimated creatinine clearance (ClCr) < 80 mL/min using Cockcroft-Gault formula

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2011-03; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Evidence of BE on single-dose pharmacokinetic parameters maximum observed concentration (Cmax) derived from Saxagliptin, 5-Hydroxy Saxagliptin and Metformin plasma concentration versus time data. | 48 hours after dosing
Evidence of BE on single-dose pharmacokinetic parameters time of maximum observed concentration (Tmax) derived from Saxagliptin, 5-Hydroxy Saxagliptin and Metformin plasma concentration versus time data. | 48 hours after dosing
Evidence of BE on single-dose pharmacokinetic parameters (AUC(0-T) derived from Saxagliptin, 5-Hydroxy Saxagliptin and Metformin plasma concentration versus time data. | 48 hours after dosing
  Area under the concentration-time curve from time zero to the time of the last quantifiable concentration (AUC(0-T))
Evidence of BE on single-dose pharmacokinetic parameters area under the concentration-time curve from time zero extrapolated to infinite time (AUC(INF)) derived from Saxagliptin, 5-Hydroxy Saxagliptin and Metformin plasma concentration versus time data. | 48 hours after dosing
Evidence of BE on single-dose pharmacokinetic parameters half-life (T-HALF) derived from Saxagliptin, 5-Hydroxy Saxagliptin and Metformin plasma concentration versus time data. | 48 hours after dosing

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 3 days after dosing
Active metabolite of Saxagliptin, 5-Hydroxy Saxagliptin, from 5 mg Saxagliptin/500 mg Metformin XR FDC tablet & from 5 mg Onglyza administered together with 500 mg Glifage® XR in single-dose fed & fasted state pharmacokinetics in healthy subjects | 3 days after dosing
  Amount of the active metabolite of Saxagliptin, 5-Hydroxy Saxagliptin (BMS-510849), from the 5 mg Saxagliptin/500 mg Metformin XR FDC tablet and from 5 mg Onglyza™ administered together with 500 mg Glifage® XR (marketed in Brazil by Merck S.A.) in single-dose fed and fasted state pharmacokinetics in healthy subjects

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Campinas, São Paulo, Brazil

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx